CLINICAL TRIAL: NCT03035526
Title: Do Endogenous Sex Hormones Affect Pericardial Adipose Tissue Volume of Males in The Multi-Ethnic Study of Atherosclerosis (MESA)?
Brief Title: Sex Hormones and Pericardial Adipose Tissue
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Aydogan Aydogdu, MD, Gulhane School of Medicine
Other Study IDs: AA1972
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Pericardial Adipose Tissue and Sex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3161 men (45-84 years old): 3161 men without known coronary artery disease

SUMMARY:
In this study, our aim is to show the relation between sex hormones and PAT and to confirm whether PAT is associated with coronary artery calcification (CAC) in different testosterone levels in the males.

ELIGIBILITY:
Inclusion Criteria:

* 3213 males
* African American
* Caucasian
* Asian (largely Chinese) and Hispanic adults aged 45-84 years and free of known cardiovascular disease at baseline (2000-2002)

Exclusion Criteria:

* Patients with known coronary artery disease

Ages: 45 Years to 84 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3161 men (45-84 years old; white, black, Hispanic, or Chinese) at 6 centers in the United States
Sampling Method: Probability Sample
Enrollment: 3213 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Relation ship between pericardial adipose tissue and sex hormones in males | years
  Total testosterone and sex hormone binding globulin levels were related with pericardial adipose tissue